CLINICAL TRIAL: NCT06821958
Title: Amplitude-modulated Radiofrequency Electromagnetic Field Treatment for Advanced Hepatocellular Carcinoma (Immune-RF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Pirus Ghadjar, Prof. Dr., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immune-RF
Record Dates: First submitted 2024-12-21; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Routine double immune checkpoint inhibition (HIMALAYA phase III trail, STRIDE-arm) combined with radiofrequency electromagnetic field treatment for 60 minutes twice a week
  Interventions: Device: Radiofrequency electromagnetic field treatment

INTERVENTIONS:
Device: Radiofrequency electromagnetic field treatment — Radiofrequency electromagnetic field treatment using a carrier frequency of 13.56 MHz

SUMMARY:
Combined double immune checkpoint inhibition and radiofrequency electromagnetic field treatment for patients with advanced hepatocellular carcinoma

DETAILED DESCRIPTION:
Charité University Medicine Berlin is currently the only German University Hospital with an available capacitive radiofrequency electromagnetic field treatment device. While there is retrospective data available regarding the assumed effectiveness and low toxicity profile of radiofrequency electromagnetic field treatment for various solid tumors including liver cancer, there is no prospective data available on the combined effect of first-line palliative double immune checkpoint inhibition and radiofrequency electromagnetic field treatment for patients with advanced hepatocellular carcinoma. The investigators aim to conduct a feasibility trial and plan to compare the results with data of a prospective trial with a comparable patient population who received double immune checkpoint inhibition alone.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with combined Anti-PD-L1 and Anti-CTLA-4 antibodies
* Written informed consent prior to any study procedure
* 18 years or older
* Histologically confirmed HCC
* HCC not amenable to curative (including resection or ablation) or locoregional (including TACE) therapies
* No prior systemic therapy for HCC
* Compensated liver function, as defined by a Child-Pugh score ≤ B7
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Measurable disease by Response Criteria in Solid Tumors (mRECIST and RECIST v1.1) criteria
* Body weight of > 30 kg
* Women of childbearing potential with negative pregnancy test and agreement for adequate birth control if conception is possible
* If present HBV and HCV managed according to the local institutional practice

Exclusion criteria:

* Arterioembolic event including a stroke or myocardial infarction within 3 months prior to randomization Severe / unstable angina, or symptomatic congestive heart failure as defined by NYHA III/IV
* Cardiac pacemakers / ICD
* Large metal implants in the treatment area
* Current evidence of coagulopathy or bleeding diathesis
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Decompensated liver function as defined by Child Pugh ≥ B8
* Patients on a liver transplantation list
* Patients with autoimmune disorders or history of organ transplantation who require immunosuppressive therapy
* Uncontrolled autoimmune or inflammatory disorders
* Patient not able for supine positioning (e.g. due to pain)
* Significantly altered mental status
* Pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Every 10-12 weeks until progression or a maximum follow-up of 3 years
  Objective response rate

SECONDARY OUTCOMES:
Acute and late toxicity | During 4 years of trial conduction
  CTCAE version 5
Quality of life (QoL) | During 4 years of trial conduction
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30
Quality of life (QoL) | During 4 years of trial conduction
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-HCC18
Progression-free survival (PFS) | During 4 years of trial conduction
  Progression-free survival
Overall survival (OS) | During 4 years of trial conduction
  Overall survival
Time to progression (TTP) | During 4 years of trial conduction
  Time to progression
Duration of response (DOR) | During 4 years of trial conduction
  Duration of response

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided